CLINICAL TRIAL: NCT05582980
Title: Online High-definition Transcranial Direct Current Stimulation Over the Left Dorsolateral Prefrontal Cortex During a Working Memory Task for Treating Negative Symptoms of Schizophrenia
Brief Title: Online HD-tDCS Over the Left DLPFC During a Working Memory Task for Treating Negative Symptoms of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Hsin-An Chang, MD, Professor, Attending Psychiatrist, Department of Psychiatry, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-108-03-002
Record Dates: First submitted 2022-10-14; First posted 2022-10-17 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder, Mixed Type; Negative Symptoms in Schizophrenia
Keywords: Schizophrenia; Negative Symptoms; Dorsolateral prefrontal cortex; HD-tDCS; Working memory tasks
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation concealment was further ensured by the administration of HD-tDCS using "study mode of the device" in which a five-digit numerical code specific to individual participant was entered into the device (Eldith DC stimulator Plus, NeuroConn, Ilmenau, Germany) that resulted in either active or sham stimulation, i.e., the researcher got the randomization code and a unique five-digit numerical code for an individual participant from the study coordinator while HD-tDCS administrator entered the code for study mode into the device. The study coordinator had continuous access to the randomization list and unblinded the study after the final visit of the last participant. Not until the unblinding of the trial did the participants, HD-tDCS administrators, researchers and clinical raters know the actual stimulation types.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HD-tDCS (active) (Experimental): Stimulation will be applied by a battery-operated device (NeuroConn DC Stimulator Plus) via 5 carbon rubber electrodes (1 cm radius, high-definition 4 × 1 rings configuration). To target the left DLPFC, the central electrode (anode) will be placed over International 10-20 electrode position F3, with return peripheral electrodes at Fp1, Fz, C3 and F7. Stimulation will be applied at an intensity of 2 milliamp (mA), 8-sec fade in and 5-sec fade out, for 20 min, two times daily, on 5 consecutive weekdays (total 10 sessions). During each session, the subject has to perform a computerized working memory task (i.e., 2-back task). The two times daily sessions will be separated by at least 2 hours.
  Interventions: Device: HD-tDCS
- HD-tDCS (sham) (Sham Comparator): In sham stimulation, the electrode montage and protocol will be the same as the active stimulation, except the 2 mA current will be turned on for 30 sec and then ramped down to 0 mA through the remainder of the 20-min time.
  Interventions: Device: HD-tDCS

INTERVENTIONS:
Device: HD-tDCS — See detail in arm/group descriptions regarding the intervention.

SUMMARY:
In this randomized double-blind trial, the investigators aim to investigate whether online high definition transcranial direct current stimulation (HD-tDCS) over the left dorsolateral prefrontal cortex (DLPFC) during a working memory task improves the severity of negative symptoms in schizophrenia patients with predominant negative symptoms.

DETAILED DESCRIPTION:
Positive (delusions and hallucinations) and negative (blunted affect, avolition-apathy, alogia and anhedonia-asociality) symptoms are recognized as core features of schizophrenia. Antipsychotic medications as the first-line treatment for schizophrenia can reduce the positive symptoms within 14-28 days but good evidence that antipsychotics have any beneficial effect on negative symptoms is scarce. Negative symptoms remain the most important unmet therapeutic needs in schizophrenia.

Accumulating functional neuroimaging research has linked the correlation between negative symptoms and reduced dorsolateral prefrontal activity. Atypical antipsychotics, the mainstream treatment for schizophrenia, are known to show little effect on patients' hypofrontality and some of them (e.g., strong dopamine receptor antagonists and clozapine) are even associated with a decrease in prefrontal activation. All these findings have driven the development of novel and effective treatments targeting the brain regions implicated in negative symptoms of schizophrenia, e.g., non-invasive brain stimulation (NIBS) of over the left DLPFC.

Transcranial direct current stimulation (tDCS) is a NIBS that has great potential to improve negative symptoms of schizophrenia. tDCS applies a weak direct current on the scalp and through the brain and rapidly leads to changes in cortical excitability by shifting membrane resting potentials, which facilitates either depolarization or hyperpolarization of the brain neurons. Repetitive stimulation during specific time intervals further enhances efficacy and prolongs the after-effects of tDCS through modifying the efficacy of N-methyl-D-aspartate receptor. An increasing number of studies attempted to reduce negative symptoms of schizophrenia by using tDCS.

Most tDCS research delivers direct current to the participants while they are at rest (offline tDCS). There has been a novel stimulation model called "online" stimulation, in which non-invasive brain stimulation is applied while the individuals are concurrently engaged in a neuropsychological task. For example, a cognitive task has been known to activate a specific brain region (e.g., working memory task and prefrontal cortex). The susceptibility of a specific brain region (i.e., prefrontal cortex) to neuro-stimulation will be enhanced if it is simultaneously activated when engaging a working memory task. Compared to the use of tDCS while the subject is at rest (offline tDCS), the application of tDCS to activate the prefrontal cortex while the subject is engaged in a working memory task (online tDCS) can potentially result in resonated effects and further enhance the neuromodulation on the target brain region, aka functional targeting.

High definition tDCS (HD-tDCS) targets cortical areas using arrays of electrodes on the scalp (i.e. a classic 4 × 1 ring configuration) and constrains the electrical current flow to a specific cortical area, allows for more accurate definition of the current field distribution than conventional tDCS and serves to optimize electrode montage to specifically target the brain areas of interest.

Our proof-of-concept study aims to investigate the efficacy of online HD-tDCS over left DLPFC as an add-on therapy to improve negative symptoms severity in schizophrenia patients with predominant negative symptoms. Moreover, it provides data on other secondary outcomes and preliminary neurophysiological data for this intervention condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 20-65 years and diagnosed with the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition ( DSM-5 ) schizophrenia or schizoaffective disorder
* Duration of illness≧1 year
* With a clinical presentation of predominant negative symptoms (according to the clinical judgment of 2 experienced psychiatrists) and the Positive and Negative Syndrome Scale (PANSS) score > 70
* Receiving stable antipsychotic drug regimen >8 weeks.

Exclusion Criteria:

* Subjects with current psychiatric comorbidity or active substance use disorder with the exception of caffeine and/or tobacco
* Having contraindications for tDCS, e.g., implanted brain medical devices or metal in the head
* Pregnancy at enrollment
* Having a history of seizures, intracranial neoplasms or surgery, severe head injuries, or cerebrovascular diseases

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The change over time in the Chinese version of the Positive and Negative Syndrome Scale Factor Score for Negative Symptoms (PANSS-FSNS) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  PANSS is a clinician-administered rating scale to measure the severity of psychopathological symptoms of the patients with schizophrenia spectrum disorder. The patient is rated from 1 to 7 on 30 different symptom items. All items scores are summed up to yield a total PANSS score, which ranges from 30 to 210. A higher score indicates greater psychopathological symptom severity. The five-factor PANSS model can be obtained by calculating from 26 of 30 items of PANSS to represent positive, negative, grandiosity/excitement, disorganization, and depression factor scores, respectively. In this model, PANSS-FSNS (7 items, N1+N2+N3+N4+N6+G7+G16, score 7-49) is selected as the primary outcome.

SECONDARY OUTCOMES:
The change over time in the score of the Chinese version of the Scale for the Assessment of Negative Symptoms (SANS) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  The Scale for the Assessment of Negative Symptoms (SANS) is used to assess negative symptoms in schizophrenia on a 25 item, 6-point scale. The SANS measures five domains of the negative symptoms including affective flattening or blunting, alogia, avolition - apathy, anhedonia - Asociality, Attention. In each domain, separate symptoms are rated from 0 (absent) to 5 (severe). A total SANS score ranges from 0 to 125.
The change over time in the scores of two subdomains of PANSS negative symptoms (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  PANSS is a clinician-administered rating scale to measure the severity of psychopathological symptoms of the patients with schizophrenia spectrum disorder, ranging from 30 to 210. A higher score indicates greater psychopathological symptom severity. Two subdomains of negative symptoms were identified from the PANSS: the Expressive Deficit domain (EXP domain, the sum of items of N1, N3, N6, G5, G7 and G13) including features of blunted affect and alogia and the Avolition-Apathy domain (AA domain, the sum of items of N2, N4, and G16) including manifestations of anhedonia, asociality and avolition.
The change over time in the scores of the five-factor PANSS model other than FSNS (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  PANSS is a clinician-administered rating scale to measure the severity of psychopathological symptoms of the patients with schizophrenia spectrum disorder, ranging from 30 to 210. A higher score indicates greater psychopathological symptom severity. The scores of five-factor PANSS model other than FSNS can be obtained by calculating from 26 of 30 items of PANSS: positive (5 items, P1+P3+P5+P6+G9,score 5-35), grandiosity/excitement (4 items, score 4-28), disorganization (5 items, score 5-35), and depression (4 items, score 4-28) factor scores.
The change over time in the score of the Chinese version of the Personal and Social Performance scale (PSP) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  A clinician-administered rating scale to measure the psychosocial functioning of the patients with schizophrenia spectrum disorder. The PSP scale measures psychosocial functioning within four domains: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior.The patient is rated from 1 to 6 on each item of the four domains. A higher score indicates greater psychosocial functioning in any of the four domains.
  The final global score is defined according to a summary instruction table. This scale provides a single, overall rating from 1 to 100, where a higher score represents better personal and social function.
The change over time in the score of the self-reported version of the graphic personal and social performance scale (SRG-PSP) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  The SRG-PSP is a self-rating scale of proven validity and reliability, comprising both male and female versions of cartoon-like pictures that are derived from the narrative text of the four domains of Personal and Social Performance (PSP) scale including the sub-items of socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behaviour.
The change over time in the score of the abbreviated version of the Scale to Assess Unawareness in Mental Disorder in schizophrenia (SUMD) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  An expert-rating scale based on a patient interview to measure patients' clinical insight. The abbreviated version of SUMD comprises 9 items measuring current states of awareness as follows: (1) a mental disorder, (2) consequences of a mental disorder, (3) effects of drugs, (4) hallucinatory experiences, (5) delusional ideas, (6) disorganized thoughts, (7) blunted affect, (8) anhedonia, and (9) lack of sociability. Scores on each item range from 0 to 3. A score of 0 indicates 'not applicable'; 1, 'aware'; 2, 'somewhat aware/unaware' and 3, 'severely unaware.' Based on the 3 dimensions approach of the abbreviated version of SUMD, the scores on the items 1-3, 4-6 and 7-9 were averaged to obtain the dimension score of 'awareness of the disease', 'awareness of positive symptoms', and 'awareness of negative symptoms', respectively. All dimension scores were linearized on a 0-100 scale, with 0 and 100 indicating the lowest and highest level of unawareness, respectively.
The change over time in the score of the Taiwanese version of the Beck Cognitive Insight Scale (BCIS) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  Cognitive insight was measured by the Taiwanese version of the Beck Cognitive Insight Scale (BCIS), a self-reported instrument comprising 15 items.The Taiwanese BCIS is composed of 2 subscales including reflective attitude (9 items) and certain attitude (6 items). We obtained a R-C (reflective attitude minus certain attitude) index of the Taiwanese BCIS, representing the measurement of cognitive insight by subtracting the score of the certain attitude subscale from that of the reflective attitude subscale. Lower R-C index scores indicate poorer cognitive insight.
The change over time in the score of the Taiwanese version of the Self-Appraisal of Illness Questionnaire (SAIQ) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  The Taiwanese version of the Self-Appraisal of Illness Questionnaire (SAIQ) was used to assess attitudes toward mental illness and experience of psychiatric treatment.This self-administered tool was composed of 17 items. The patients rated the extent to which they agreed with each statement of the item by using a four-point Likert scale, ranging from 1, ''do not agree at all'', to 4, ''completely agree''. Whether the scale score is in order from least to most or from the most to least depends on the content of the item statement. The total score of SAIQ ranges from 17 to 68.
The change over time in the score of the Chinese version of the Schizophrenia Quality of Life Scale Revision Four (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  The Chinese version of the Schizophrenia Quality of Life Scale Revision Four is a self-administered questionnaire of 33 items in two domains: psychosocial and vitality. All but four items are coded on a scale of 0-4 according to the frequency of occurrence during the previous 7 days (0 = always, 4 = never; the four exceptions are coded 0 = never, 4
  = always). A higher score indicates higher health-related QoL.
The change over time in the scores of Taiwanese version of Medication Adherence Rating Scale (from baseline to the timepoints immediately after intervention and at one-week follow-up). | Two weeks
  The Taiwanese version of Medication Adherence Rating Scale (MARS), translated from the original MARS, was used to assess patients' beliefs about medication adherence. The translated MARS contains 10 yes/no items. Items 1-5 form the medication adherence subscale and items 6-10 form the subjective response to taking medication subscale. The scores from MARS subscales are summed to yield a total MARS score ranging from 0 (poor adherence to treatment) to 10 (good adherence to treatment), indicating a broad measure of medication compliance.
The change over time in the total score of the Extrapyramidal Symptoms Rating Scale (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  Extrapyramidal Symptoms Rating Scale (ESRS) is a quantitative measure of antipsychotic-induced extrapyramidal movement symptoms. The ESRS is composed of the patient-assessed ESRS questionnaire and the physician-rated subscales for assessing parkinsonism/akathisia, dystonia movement, and dyskinesia movement.
The changes over time in the results of Digit span (forward and backward) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  A test to measure the capacity of working memory of the patients
The changes over time in the results of Finger tapping test (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  A neuropsychological test that examines motor functioning, specifically, motor speed and lateralized coordination.
The changes over time in the results of Continuous Performance (CPT, version 2.0) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  A neuropsychological test that examines the performance of prefrontal-mediated task.
The changes over time in the results of Wisconsin Card Sorting Test (WCST) (from baseline to the timepoints immediately after intervention and at one-week follow-up). | Two weeks
  A neuropsychological test of "set-shifting", i.e. the ability to display flexibility in the face of changing schedules of reinforcement.
The changes over time in the results of Tower of London test (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  A neuropsychological test for the assessment of executive functioning specifically to detect deficits in planning, which may occur due to a variety of medical and neuropsychiatric conditions.
The changes over time in the results of Color Trails Test (CTT) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  The CTT, a culture-neutral version of the Trail Making Test, was selected to measure sustained visual attention. The CTT consists of two parts (CTT-1 and CTT-2). The CTT-1 requires participants to connect a series of numbered circles that are randomly printed on a sheet of paper. In the CTT-2, numbered circles of 1 to 25 are shown twice (printed in pink and in yellow) randomly on a sheet of paper. Participants are asked to connect the numbers from 1 to 25 alternating between the two colors.
The changes over time in the results of Stroop Color Word Test (SCWT) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  Stroop Color Word Test (SCWT), Chinese version; was administered to measure selective attention and cognitive flexibility. SCWT is composed of three parts, each lasting for 45 seconds.
The changes over time in indices of heart rate variability (HRV) measured at baseline, the end of stimulation, and 1-week follow-up. | Two weeks
  HRV indices represent autonomic functioning. ECG electrodes were placed on bilateral arms just below the elbows, with a ground electrode placed just above the right wrist bone. Lead I electrocardiogram of each patient was taken for 5 min after sitting and having a rest for 20 min in a soundproof, dim-lighted room with thermostatic control. At the four timepoints (baseline, after 10-session HD-tDCS, at 1-week and 1-month follow-ups), HRV will be collected during resting and during a dual 2-back task. The ECG signals were acquired, stored, pre-processed according to the recommended procedures and processed by an HRV analyser (LR8Z11, Yangyin Corp., Taipei, Taiwan). The time domain of HRV is obtained: Standard deviation of NN intervals (SDNN). Power spectrum of HRV is quantified into the standard frequency-domain measurements including low-frequency power (LF, 0.04-0.15 Hz), high-frequency power (HF, 0.15- 0.40 Hz).
The changes over time in EEG absolute power and lag phase synchronization in the frontal electrodes in the delta, theta, alpha, beta and gamma range (from baseline to the end of stimulation). | One week
  In a recliner in a dimly lit, electrically shielded room, patients' EEGs were recorded at baseline and at the end of stimulation by using the Neuro Prax® TMS/tDCS full-band DC-EEG system with 32 EEG Ag/AgCl electrodes in the standard 10-20 International placement. EEG will be collected with eye opened (5min) and closed (5min). Signals will be amplified in the dynamic input range of ± 140 mV at a resolution of 0.5 μV by using EEG amplifiers and stored for offline analyses. Eye or muscle artifacts were automatically detected and removed using NeuroPrax's built-in software.
The changes over time in high density near infrared spectroscopy (from baseline to the end of stimulation). | One week
  Cognitive task protocol used for the functional near infrared spectroscopy (fNIRS) system to measure the relative changes in oxy Hb and deoxy Hb. Hemoglobin Hb changes will be measured during 2 different cognitive tasks: semantic verbal fluency task (SVFT) and and a 2 back task . An SVFT involves generating as many words as possible within a certain time frame and hints at the semantic category of the words generated. The task measures the amount of information regarding categorization and the number of words that can be retrieved from memory in 1 min. The task involved generating as many words as possible in relation to the keywords. The 2 back task is used to evaluate participants' working memory. The examiner presents the words while the participant performs the working memory, and the number of memorized words is measured afterward. In this task, participants de

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-An Chang, M.D., Principal Investigator — Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan
Locations (1):
- Tri-service general hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma CC, Lin YY, Chung YA, Park SY, Huang CC, Chang WC, Chang HA. The two-back task leads to activity in the left dorsolateral prefrontal cortex in schizophrenia patients with predominant negative symptoms: a fNIRS study and its implication for tDCS. Exp Brain Res. 2024 Mar;242(3):585-597. doi: 10.1007/s00221-023-06769-5. Epub 2024 Jan 16. PMID 38227007